CLINICAL TRIAL: NCT01999725
Title: A Randomized, Double-Blind, Placebo-Controlled, Ascending One-Day (Single and Divided Dose) Safety, Tolerability, and Pharmacokinetic Study of EDP-788 in Healthy Adult Volunteers
Brief Title: Evaluation of the Safety and Pharmacokinetics of a Single Oral Dose of EDP-788
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Enanta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDP788-001
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2015-01-09 (Estimated); Status verified 2015-01

CONDITIONS: Safety in Normal Volunteers
Keywords: Normal Volunteers, Safety, Pharmacokinetics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EDP-788 (Experimental): Single doses with dose escalation to continue in successive cohorts
  Interventions: Drug: EDP-788
- Placebo (Placebo Comparator): Single dose with matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: EDP-788 — EDP-788 Capsules and matching placebo capsules. EDP-788 Liquid Suspension and matching placebo. All interventions are given as single doses
  Arms: EDP-788
Drug: Placebo — Matching placebo capsules or matching suspension
  Arms: Placebo

SUMMARY:
The primary objective of the study is to determine the safety of single doses of orally administered EDP-788.

Secondary objectives of the study are:

* To describe the pharmacokinetics of EDP-788 (and its metabolite EDP-322) after single doses of orally administered drug
* To estimate the bioavailability of EDP-788 capsules relative to an oral liquid suspension
* To estimate the effect of co-administration of food on the absorption of EDP-788

DETAILED DESCRIPTION:
Subjects are enrolled in successive cohorts and are randomized to receive either EDP-788 or placebo capsules. If the safety profile of the drug is acceptable, based upon review of blinded data, the cohort receiving the next higher dose will be treated. Up to 8 cohorts will be recruited. All subjects receive a single dose of study drug (EDP-788 or placebo).

Subjects in Cohort C will receive a second single dose of study drug (EDP-788 or placebo) approximately 2 weeks after the first dose. The second dose will be administered as a liquid suspension rather than as a capsule formulation. The purpose of the second dose is to estimate the bioavailability of the capsule formulation relative to the suspension.

Subjects in Cohort E will receive a second single dose of study drug (EDP-788 or placebo) approximately 2 weeks after the first does. The second dose will be administered with a standard test meal. The purpose of the second dose is to estimate the effect of food on absorption of EDP-788.

ELIGIBILITY:
Key Inclusion Criteria:

* In good general health
* BMI between 18 - 32 kg/m2
* Women must be of non-childbearing potential (surgically sterilized)
* Normal electrocardiogram
* Willing to abstain from strenuous physical exercise starting 3 days prior to admission to the study clinic through the 8 - 10 day post-dosing visit

Key Exclusion Criteria:

* Hypersensitivity to macrolide antibiotics
* Abnormal laboratory values
* History of gastrointestinal surgery which may interfere with drug absorption
* Active Hepatitis B, Hepatitis C, or HIV infection
* Use of prescription or non-prescription drugs within 14 days of study drug administration
* Use of nicotine within 3 months of study drug administration

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | From time of dosing to 8 - 10 days after receiving study drug

SECONDARY OUTCOMES:
Changes from baseline in laboratory values and vital signs | From time of dosing to 8 - 10 days after receiving study drug

OTHER OUTCOMES:
Pharmacokinetic parameters | From time of dosing to 3 days after receiving study drug

CONTACTS AND LOCATIONS:
Overall Officials: Theresa T Pham, MD, Principal Investigator — PPD Phase I Clinic
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States